CLINICAL TRIAL: NCT06493448
Title: Prospective Observational Study of Gastric Cancer Synchronous Liver Metastases: a Multi-centre, Noninterventional, Cohort Study
Brief Title: Prospective Observational Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Lin Chen (Other)
Collaborators: Peking University International Hospital (Other); Chinese PLA General Hospital (Other)
Responsible Party: Sponsor-Investigator, Lin Chen, Director and Clinical Professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: XHongqing
Record Dates: First submitted 2024-04-22; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Gastric Cancer; Liver Metastases
Keywords: gastric cancer; liver metastasis; observation; treatment; prognosis
MeSH Terms: conditions — Stomach Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort A: Type I liver metastases, resectable type, with the option of direct surgical resection or preoperative systemic therapy
  Interventions: Other: observation
- Cohort B: Type II liver metastases, potentially resectable type, preoperative systemic therapy is applied to gain the chance of surgery
  Interventions: Other: observation
- Cohort C: Type III liver metastases, systemic treatment according to recommended guidelines and patient characteristics
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — This is an observational study.

SUMMARY:
The goal of this observational study is to learn about the overall disease status, diagnostic and therapeutic modalities, and prognosis of patients with gastric cancer liver metastasis(GCLM) in China. The investigators divided the participants into three groups( three types) of gastric cancer liver metastasis based onChinese c-GCLM classification system.The main question it aims to answer is:

1. How long do patients with GCLM live?
2. How different treatment modalities (surgery, chemotherapy, immunotherapy, targeted therapy and others) affect patients' prognosis of three type? All participants will be tracked for their physical condition.

DETAILED DESCRIPTION:
This is a prospective, non-interventional, observational, multi-centre, real-world study designed to monitor the general condition, treatment pattern and prognosis of patients with GCLM. GCLM patients were divided into 3 types: Type I (resectable type), Type II (potentially resectable type), Type III (unresectable type). The patients' general information, past medical history, imaging results, laboratory tests, surgical and systemic therapy details will be recorded and analysed. The 2-year overall survival (OS) will be recorded as the primary endpoint. The different therapies (surgery, chemotherapy and immunotherapy) of GCLM, the effects of different therapies on prognosis including OS of type I, II and III; R0 resection rate and diease free survival (DFS) of type I; successful conversion rate and R0 resection rate and events free survival (EFS) of type II will be recorded as secondary endpoints.

This study involving human participants were reviewed and approved by the Ethics Committee of Chinese PLA General Hospital (No.S2023-724-02) and will be conducted according to the guidelines of the Declaration of Helsinki. Study findings will be disseminated through international peer-reviewed journal articles as well as public, academic presentations at national and international conferences.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years
* gastric primary lesions confirmed by pathology and liver metastases confirmed by pathology or imaging (before, during, or after initial treatment)
* expected survival time of ≥ 12 weeks
* Eastern Cooperative Oncology Group Physical Status Score (ECOG PS score) of 0-2
* signed informed consent
* good compliance and ability to complete regular follow-up

Exclusion Criteria:

* heterochronous liver metastases
* multi-centra clinics with significant missing case information
* diagnosed, suspected or active autoimmune disease
* history of immunodeficiency
* history of allogeneic organ and haematopoietic stem cell transplantation
* pregnant or breastfeeding female patients
* uncontrolled co-morbidities, including but not limited to:
* a.HIV-infected (HIV-positive) patients
* b.severe infections that are active or poorly controlled clinically
* c.evidence of severe or uncontrolled systemic disease
* - severe psychiatric disease
* - severe neurological disease
* - epilepsy
* - dementia
* - unstable or uncompensated respiratory
* - cardiovascular
* - hepatic disease
* - renal disease
* - uncontrolled hypertension
* Abnormal coagulation in people with active bleeding or new thrombotic disease, on therapeutic doses of anticoagulants, or with bleeding tendencies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The main study population was: patients diagnosed with liver metastases from gastric cancer who met the inclusion and exclusion criteria in China. Patient care in various tertiary hospitals throughout the country.
Sampling Method: Non-Probability Sample
Enrollment: 1326 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year OS | 2 years OS from diagnosed time to measured time or death
  The primary study endpoint was two-year survival in patients

SECONDARY OUTCOMES:
OS of type I（questionnaires, phone calls, and outpatient follow-up.） | OS from diagnosed time to measured time or death（up to 5 years）
  the effects of different therapeutic modalities (surgery, chemotherapy, immunotherapy, targeted therapy and others) on prognosis.
OS of type II （questionnaires, phone calls, and outpatient follow-up.） | OS from diagnosed time to measured time or death（2 to 5 years）
  the effects of different therapeutic modalities (surgery, chemotherapy, immunotherapy, targeted therapy and others) on prognosis.
OS of type III（questionnaires, phone calls, and outpatient follow-up.） | OS from diagnosed time to measured time or death（no more than 2 years）
  the effects of different therapeutic modalities (surgery, chemotherapy, immunotherapy, targeted therapy and others) on prognosis.
DFS of type I（questionnaires, phone calls, and outpatient follow-up.） | Through study completion, an average of 2 year.
  DFS of type I. Disease-free survival time maintained after the participant has been saved by therapeutic measures.Especially in patients underwent radical surgery.
R0 resection rate (pathological information from medical record.) | Through study completion, an average of 2 year.
  Proportion of all operated patients achieving radical resection.
successful conversion therapy rate (pathological information and surgery information from medical record.) | Through study completion, an average of 2 year.
  Proportion of type II patients underwent radical surgery after systemic treatment.

OTHER OUTCOMES:
Objective response rate (ORR) of disease by immunological drugs (Imaging information, pathology information from medical record.) | Through study completion, an average of 2 year.
  Degree of tumour response after treatment in all participants treated with applied immunological drugs.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lu T, Gao Y, Zhang G, Zhang H, Chen Z, Liu Y, Chen L, Xi H. Gastric cancer liver metastases in China: a real-world, multicentre, prospective, observational cohort study protocol. BMJ Open. 2025 Jan 8;15(1):e086276. doi: 10.1136/bmjopen-2024-086276. PMID 39779263